CLINICAL TRIAL: NCT02011997
Title: Comparison of Video-assisted Thoracoscopic Segmentectomy Versus Lobectomy for Lung Adenocarcinoma in Situ and With Microinvasion
Brief Title: Comparison of cVATS Segmentectomy Versus Lobectomy for Lung Adenocarcinoma in Situ and With Microinvasion
Acronym: cVATS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, President, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAH-GZU-001
Record Dates: First submitted 2013-11-16; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Non-small Cell Lung Cancer Stage I; Lung Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- segmentectomy (Experimental): Patients undergo cVATS (complete Video-assisted Thoracoscopic Surgery) segmentectomy
  Interventions: Procedure: patients undergo cVATS segmentectomy
- Lobectomy (Active Comparator): Patients undergo cVATS lobectomy
  Interventions: Procedure: Patients undergo cVATS lobectomy

INTERVENTIONS:
Procedure: patients undergo cVATS segmentectomy
  Arms: segmentectomy
Procedure: Patients undergo cVATS lobectomy
  Arms: Lobectomy

SUMMARY:
This is a Prospective, open-label, parallel, multi-center, Phase III randomized trial to evaluate the efficacy and safety of video-assisted thoracoscopic segmentectomy versus Lobectomy in treating patients with Lung adenocarcinoma in situ or with microinvasion.

DETAILED DESCRIPTION:
Lobectomy has long been considered the standard procedure for early-stage lung cancer, and minimally invasive techniques have been demonstrated to be associated with superior outcomes compared with lobectomy by thoracotomy. the us of segmentectomy is under investigation for selected patients with small tumors, and the use of minimally invasive strategies is applicable as well.

This nationwide, multicenter, prospective, randomized open phase III study of cVATS (complete Video-assisted Thoracoscopic Surgery) segmentectomy versus Lobectomy for stage IA non-small cell lung cancer (NSCLC) patients with Lung adenocarcinoma in situ or with microinvasion, is aiming to evaluate the relapse free survival and 5 year overall survival (OS) rate of two types of surgery. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo cVATS lobectomy.
* Arm II: Patients undergo cVATS segmentectomy.

Patients will be followed up every 3 months within the first year, and annually for 5 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Preoperative criteria: peripheral non-small cell lung cancer, no larger than 2 cm in maximal diameter, no lymph node metastasis, FEV1%>50% (FEV1: Forced Expiratory Volume in 1 second);

Preoperative imaging:pure ground-glass or mixed ground-glass nodules (part-solid, solid areas < 0.5cm);

Follow-up duration last 3 months or more, HRCT (HRCT: high-resolution computed tomography) lesion maximum diameter was measured three times and took the average, meet the criteria of clinical surgical indications;

Intraoperative criteria: histologically confirmed NSCLC, adenocarcinoma in situ or with microinvasion;

No prior ipsilateral thoracotomy;

No prior anti-neoplastic therapy;

EOCG Performance status 0-2;

Sufficient organ functions;

Written informed consent.

Exclusion Criteria:

Active bacterial or fungous infection;

Simultaneous or prior (within the past 5 years) other malignant disease;

Interstitial pneumonitis, pulmonary fibrosis, or severe COPD (COPD: chronic obstructive pulmonary disease);

Abnormal Psychosis;

Uncontrollable diabetes mellitus;

History of severe cardiovascular disease;

Any condition which, in the opinion of the investigator might interfere with the evaluation of the objective.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | From date of randomization until the date of first documented relapse or metastasis, whichever came first, assessed up to 5 years
  Compare the relapse-free survival (RFS) of patients with lung adenocarcinoma in situ or microinvasion undergoing cVATS segmentectomy vs lobectomy.

SECONDARY OUTCOMES:
5-year survival rate | participants are followed until death or up to 5 years
  Compare the 5-year survival rate of patients undergoing cVATS segmentectomy vs lobectomy
postoperative complication | 0 to 3 months postoperatively
  Compare the postoperative complication rate of patients undergoing cVATS segmentectomy vs lobectomy
pulmonary function | 6 months after surgery
  to evaluate the pulmonary function as measured by expiratory flow rate of the two groups 6 months postoperatively
Quality of Life | 0 to 6 months postoperative
  To evaluate the quality of life (QoL) of these patients, as measured by questionnaire of FACT-L (4th edition) and LCSS (Lung Cancer Symptom Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Principal Investigator — First Affiliated Hospital of Guangzhou Medical University
Locations (6):
- China (6):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital Zhejiang University colleague of Medicine, Hangzhou, Zhejiang
  - China-Japan Friendship hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - Shanghai Chest Hospital, Shanghai

REFERENCES:
- [Background] Van Schil PE, Asamura H, Rusch VW, Mitsudomi T, Tsuboi M, Brambilla E, Travis WD. Surgical implications of the new IASLC/ATS/ERS adenocarcinoma classification. Eur Respir J. 2012 Feb;39(2):478-86. doi: 10.1183/09031936.00027511. Epub 2011 Aug 4. PMID 21828029
- [Background] Ginsberg RJ, Rubinstein LV. Randomized trial of lobectomy versus limited resection for T1 N0 non-small cell lung cancer. Lung Cancer Study Group. Ann Thorac Surg. 1995 Sep;60(3):615-22; discussion 622-3. doi: 10.1016/0003-4975(95)00537-u. PMID 7677489
- [Background] Koike T, Togashi K, Shirato T, Sato S, Hirahara H, Sugawara M, Oguma F, Usuda H, Emura I. Limited resection for noninvasive bronchioloalveolar carcinoma diagnosed by intraoperative pathologic examination. Ann Thorac Surg. 2009 Oct;88(4):1106-11. doi: 10.1016/j.athoracsur.2009.06.051. PMID 19766789
- [Background] Yan TD, Black D, Bannon PG, McCaughan BC. Systematic review and meta-analysis of randomized and nonrandomized trials on safety and efficacy of video-assisted thoracic surgery lobectomy for early-stage non-small-cell lung cancer. J Clin Oncol. 2009 May 20;27(15):2553-62. doi: 10.1200/JCO.2008.18.2733. Epub 2009 Mar 16. PMID 19289625